CLINICAL TRIAL: NCT07393477
Title: Efficacy and Safety Profile of Becotatug Vedotin(EGFR-Targeting ADC) in Combination With Pucotenlimab and Cisplatin as Neoadjuvant Therapy for Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma (LA-HNSCC)
Brief Title: Neoadjuvant Becotatug Vedotin Plus Pucotenlimab and Cisplatin for Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRSH2025-2020; ChiCTR2600115972 (Registry Identifier: China Clinical Trial Registry)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Combined Modality Therapy; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Therapy with Becotatug Vedotin, Pucotenlimab, and Cisplatin (Experimental): Participants in this arm will receive a combination of Becotatug Vedotin (EGFR-Targeting ADC), Pucotenlimab (PD-1 Inhibitor), and Cisplatin as neoadjuvant therapy for locally advanced head and neck squamous cell carcinoma (LA-HNSCC). The treatment will be administered for approximately 6-12 weeks, followed by surgery. Participants will be monitored for safety and efficacy through routine check-ups and pathological assessments.
  Interventions: Combination Product: Combination Therapy with Becotatug Vedotin, Pucotenlimab, and Cisplatin

INTERVENTIONS:
Combination Product: Combination Therapy with Becotatug Vedotin, Pucotenlimab, and Cisplatin — Neoadjuvant therapy: Becotatug Vedotin 2.0mg/kg + Pucotenlimab 200mg + Cisplatin 75mg/m2, all administered via intravenous infusion on Day 1 (d1), with a 21-day treatment cycle for a total of 2-4 cycles (the exact number of cycles is determined by the investigator based on imaging findings, laryngoscopy results, etc.)

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of Becotatug Vedotin (EGFR-Targeting ADC) in combination with Pucotenlimab and Cisplatin as neoadjuvant therapy for patients with locally advanced head and neck squamous cell carcinoma (LA-HNSCC).

The primary objective is to assess whether this combination therapy improves the pathological complete response (pCR) rate and to evaluate its safety and tolerability. The secondary objective includes evaluating 1-year disease-free survival (DFS) rates and major pathological response (MPR) rates in patients treated with this combination therapy.

Main Questions This Trial Aims to Answer:

1. Does the combination of Becotatug Vedotin, Pucotenlimab, and Cisplatin lead to higher rates of pathological complete response (pCR) and major pathological response (MPR) in patients with locally advanced head and neck squamous cell carcinoma (LA-HNSCC)?
2. What are the safety and tolerability profiles of the combination therapy?
3. Does the treatment improve disease-free survival at 1 year after treatment?

What Participants Will Do:

Treatment: Participants will receive Becotatug Vedotin (EGFR-Targeting ADC), Pucotenlimab, and Cisplatin as a combination therapy in the neoadjuvant setting.

Treatment Duration: Treatment will last approximately 6-12 weeks, depending on the patient's individual regimen.

Follow-up Visits: Participants will attend routine check-ups for safety evaluations and pathological assessments approximately 7 weeks after completing neoadjuvant therapy.

Outcomes: Researchers will assess pathological complete response (pCR), major pathological response (MPR), and 1-year disease-free survival (DFS) following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years (inclusive).
2. Histopathologically confirmed Stage III/IVA head and neck squamous cell carcinoma (HNSCC) of the oropharynx, oral cavity, hypopharynx, or larynx (per 8th edition AJCC Cancer Staging Manual).
3. Measurable primary lesions per RECIST v1.1.
4. Treatment-naive (no prior anti-tumor therapy for current disease).
5. ECOG performance status 0-1.
6. Eligible for elective standard surgery plus adjuvant chemoradiotherapy/radiotherapy (investigator-assessed).
7. No active autoimmune diseases.
8. No concurrent malignant tumors.
9. Estimated life expectancy >= 6 months.
10. Available tumor tissue for PD-L1 IHC testing (22C3 DAKO assay).
11. Adequate hematological function (screening): ANC >= 1.5×10⁹/L, platelets >= 100×10⁹/L, Hb >= 100 g/L, WBC >= 3.5×10⁹/L; no blood transfusion or bleeding tendency within 7 days.
12. Normal liver function: ALT, AST, ALP, serum bilirubin <= 1.5×ULN.
13. Normal renal function: Serum Cr <= 1.5×ULN or creatinine clearance > 60 mL/min.
14. HPV status confirmed by p16 IHC and in situ hybridization (ISH).
15. Voluntary participation with signed informed consent; legal guardian-signed consent for incompetent subjects, and witness-supervised consent for illiterate subjects.

Exclusion Criteria:

1. Cachexia or multiple organ failure.
2. Active autoimmune disease of any type.
3. Concomitant second primary malignancy (e.g., esophageal cancer).
4. Severe active infection requiring systemic therapy.
5. Uncontrolled serious medical conditions interfering with study treatment (e.g., severe heart/cerebrovascular disease, uncontrolled diabetes/hypertension, active peptic ulcer).
6. Dementia, altered mental status, or other conditions impairing informed consent or questionnaire completion.
7. Peripheral neuropathy >= Grade 2 per CTCAE v5.0.
8. Hearing impairment >= Grade 2 per CTCAE v5.0.
9. History of malignancy within 5 years prior to screening.
10. Known HIV-positive status or diagnosed AIDS.
11. Nasopharyngeal carcinoma or HNSCC at sites other than oral cavity, oropharynx, larynx, hypopharynx (e.g., paranasal sinuses, unknown primary).
12. Receipt of investigational drugs or participation in other interventional trials within 30 days prior to screening.
13. Systemic glucocorticoids (>10 mg prednisone equivalent/day) or other immunosuppressants within 14 days prior to randomization (inhaled/topical steroids and adrenal hormone replacement are permitted without active autoimmune disease).
14. Pregnant/lactating women; subjects of childbearing potential refusing contraception.
15. Active infection requiring treatment or systemic anti-infective use within 1 week prior to first dose.
16. Live vaccine administration within 30 days prior to first dose.
17. Vulnerable populations (e.g., mental illness, cognitive impairment, critically ill status).
18. Other conditions deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response(pCR) Rate | Within 7 weeks after the completion of neoadjuvant therapy

SECONDARY OUTCOMES:
Major Pathological Response(MPR) Rate | Within 7 weeks after the completion of neoadjuvant therapy
1-Year Disease-Free Survival | 1 year after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China